CLINICAL TRIAL: NCT04511416
Title: Preventing Cognitive Decline with Metformin:: the MetMemory Study
Brief Title: Preventing Cognitive Decline with Metformin
Acronym: MetMemory
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Garvan Institute of Medical Research (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2020-07-02; First posted 2020-08-13 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Decline
Keywords: cognitive decline; dementia; cerebrovascular disease; insulin resistance; neurodegeneration; inflammation; diabetes
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Cerebrovascular Disorders; Insulin Resistance; Nerve Degeneration; Inflammation; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: randomised placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Metformin
  Interventions: Drug: Metformin XR, 500-2000mg nocte
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Metformin XR, 500-2000mg nocte

INTERVENTIONS:
Drug: Metformin XR, 500-2000mg nocte — Metformin XR, 500-2000mg nocte
  Other Names: Placebo

SUMMARY:
A randomised control study of metformin in people with mild cognitive impairment and without diabetes mellitus to determine effects on cognitive decline and neuroimaging over 3 years.

DETAILED DESCRIPTION:
A randomised placebo-control study of metformin in people with mild cognitive impairment and without diabetes mellitus to determine effects on cognitive decline, neuroimaging and biomarkers over 3 years.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese (body mass index >25.0 kg/m2, waist: women>80 cm, men>94cm;
* Mild cognitive impairment (Mild Neurocognitive Disorder), based on DSM-5 criteria;
* Fasting blood glucose <7.0 mmol/L and HbA1c <6.5%;
* Able to undertake neurocognitive testing in English.
* Not participating in another trial of drugs or lifestyle modification to reduce cognitive decline.

Exclusion Criteria:

* Life-threatening illnesses to preclude participation in a 3-year study;
* Contraindications to the use of metformin (severe heart failure or eGFR <40).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
changes in memory Z-score | 3 years
  memory domain Z-score, derived from the following neuropsychological tests: i. Rey Auditory Verbal Learning Test (RAVLT); ii. Total Learning and Delayed recall; iii. the Logical Memory Story A- Immediate Recall; and iv. Delayed Recall tests.
changes in executive function Z-score | 3 years
  executive function domain Z-score, derived from the following neuropsychological tests: i. Alphabet test; ii. D-KEFS Stroop; iii. Trail Making Test Part B; iv. Weschler Adult Intelligence Scale-IV (WAIS-IV) Digit Span Backward test.

SECONDARY OUTCOMES:
changes in processing speed domain Z-score | 3 years
  processing speed domain measured by the i. WAIS-IV Coding; and ii. Trail Making Test part B
changes in language performance domain Z-score | 3 years
  language performance domain measured by the Category Fluency (Animals) neuropsychological test
changes in attention performance domain Z-score | 3 years
  attention performance domain Z-score, measured by the WAIS-IV Digit Span Forward neuropsychological test
changes in Cogstate brief battery performance Z-score | 3 years
  computerised cognition testing using the on-line test, the Cogstate brief battery (CBB)
changes in total brain volume (cubic millimetres) | 3 years
  total grey and white matter volume
changes in hippocampal volume (cubic millimetres) | 3 years
  volume of the right and left hippocampal regions of the brain
changes in parahippocampal volume (cubic millimetres) | 3 years
  volume of the right and left parahippocampal regions of the brain
changes in brain white matter hyperintensity number | 3 years
  the number of white matter hyperintensities visualised in bain imaging by magnetic resonance imaging
changes in cerebral blood flow (mL / 100 g / min) | 3 years
  Cerebral blood flow will be measured using arterial spin labelling
changes in cerebral amyloid tracer standardized uptake value ratio (SUVR) | 3 years
  standardized uptake value ratio of amyloid tracer using positron emission tomography
changes in cognitive performance Z-score using the NIH tool box | 3 years
  The NIH Toolbox currently contains the following cognitive tests: Flanker, Pattern Comparison, Picture Sequence Memory and Dimensional Change Card Sort.
change in BOLD (blood-oxygen-level-dependent) time-series signals measured by functional magnetic resonance imaging | 3 years
  change blood oxygen-level-dependent time-series signals, measured by functional MRI
changes in biomarkers, including fasting glucose (mmol/L) and insulin (mIU/L), insulin resistance (HOMA-IR index) | 3 years
  fasting glucose (mmol/L) and insulin (mIU/L), insulin resistance (HOMA-IR index)

CONTACTS AND LOCATIONS:
Locations (1):
- Garvan Institute of Medical Research, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No